CLINICAL TRIAL: NCT00972582
Title: Determination of the Tolerable Upper Limit of Leucine Intake in Adult Humans
Brief Title: Upper Limit of Leucine Intake in Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr. Paul Pencharz, Emeritus Scientist, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: 1000012066
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Healthy
Keywords: leucine intake; tolerable upper limit; adults; amino acid supplements; Excessive Leucine Intake

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Leucine (Experimental)
  Interventions: Dietary Supplement: Leucine Increase

INTERVENTIONS:
Dietary Supplement: Leucine Increase — Graded stepwise increases in leucine intakes (50, 250, 500, 750, 1000, 1250 and 1500mg/kg/day)

SUMMARY:
When dietary amino acid supplements are consumed by humans they are normally in addition to their normal daily requirements. The investigators' laboratory played a leading role in defining the estimated average requirement (EAR) and the recommended dietary intake for the "essential" amino acids (Dietary Reference Intakes 2005). The other important but less well studied component of Dietary Reference Intakes (DRI) is - What is a safe upper limit of intake? The investigators now propose to determine the safe upper limits of the dietary essential amino acids. The recently published DRI (2005) defines the Tolerable Upper Intake Level (UL) as 'the highest average daily nutrient intake level that is likely to pose no risk of adverse health effects to almost all individuals in the general population.' As intake increases above the UL, the potential risk of adverse effects may increase'. In this proposal, the investigators define a novel method to define the safe upper limit where the 'maximum oxidative potential' of an amino acid identifies the 'metabolic limit' to dispose the amino acid. Intakes of amino acid above this level will increase the potential for adverse effects to appear.

DETAILED DESCRIPTION:
The objective of the study will be to determine the 'metabolic limit' of leucine oxidation in healthy young men by:

A) Measuring leucine oxidation in response to short term (8 hr) graded excess leucine intake B) Correlating changes in leucine oxidation with changes in plasma concentrations of keto-isocaproic acid (KIC, the first breakdown product of leucine metabolism), other essential amino acids, ammonia, urea, creatinine, glucose, insulin, and electrolytes (sodium, potassium, chloride) to identify potential biomarkers C) Correlating changes in leucine oxidation with changes in urinary excretion of leucine and ketoisocaproic acid (KIC), urea and creatinine to identify potential biomarkers

ELIGIBILITY:
Inclusion Criteria:

* Male
* 18-35 years old

Exclusion Criteria:

* Report a recent history of sudden weight loss
* Have unusual dietary habits such as chronic consumption of caffeinated beverages or alcohol
* Have any endocrine disorders
* Are currently using any prescribed medications

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Breath carbon dioxide production | Study Visits 1-7 (-45min,-30min,-15min, +2.5hrs, +3hrs, +3.5Hrs +4hrs)

SECONDARY OUTCOMES:
Plasma | Study Visits 1-7 (Hourly)
Urine | Study Visits 1-7 (8hr timepoint)
VCO2 | Study Visits 1-7 (after 5hr meal)

CONTACTS AND LOCATIONS:
Overall Officials: Paul B Pencharz, MD, Principal Investigator — The Hospital for Sick Children, Toronto, Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Elango R, Chapman K, Rafii M, Ball RO, Pencharz PB. Determination of the tolerable upper intake level of leucine in acute dietary studies in young men. Am J Clin Nutr. 2012 Oct;96(4):759-67. doi: 10.3945/ajcn.111.024471. Epub 2012 Sep 5. PMID 22952178